CLINICAL TRIAL: NCT04129515
Title: Phase I and II Study of NovoTTF-200A and Pembrolizumab in Newly Diagnosed Melanoma Brain Metastasis
Brief Title: NovoTTF-200A + Pembrolizumab In Melanoma Brain Metastasis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Contract Issues
Sponsor: Brown University (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 416
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Melanoma; Melanoma Brain Metastasis
Keywords: Melanoma Brain Metastasis; Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PHASE 1: NovoTTF-200A + PEMBROLIZUMAB (Experimental): The Phase I portion of the study will have a 3 + 3 design and consist of one cohort treated
  * NovoTTF-200A will be applied continuously, with 21 consecutive days defined as a treatment cycle.
  * Pembrolizumab will be administered once every 3 weeks, with 21 consecutive days also defined as a treatment cycle
  Interventions: Device: NovoTTF-200A; Drug: Pembrolizumab
- PHASE 2: NovoTTF-200A + PEMBROLIZUMAB (Experimental): * NovoTTF-200A will be applied continuously, with 21 consecutive days defined as a treatment cycle.
  * Pembrolizumab will be administered once every 3 weeks, with 21 consecutive days also defined as a treatment cycle
  Interventions: Device: NovoTTF-200A; Drug: Pembrolizumab

INTERVENTIONS:
Device: NovoTTF-200A — •NovoTTF-200A will be applied continuously, with 21 consecutive days defined as a treatment cycle
Drug: Pembrolizumab — Pembrolizumab will be administered once every 3 weeks, with 21 consecutive days also defined as a treatment cycle
  Other Names: Keytruda®

SUMMARY:
This research study involves studying a device as a possible treatment for metastatic melanoma in the brain. The purpose of this study is to obtain information on the safety and effectiveness of the study device, NovoTTF-200A, in melanoma participants with brain metastases when it is combined with Pembrolizumab.

The name of the study device involved in this study is:

-- NovoTTF-200A

The name of the drug used in this study is:

-- Pembrolizumab

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* The name of the study device involved in this study is: NovoTTF-200A
* The name of the drug used in this study is: Pembrolizumab
* Eligible participants will be in this research study for up to 2 years, or until progressive disease or unacceptable toxicity as is reflected in the protocol.
* This is a Phase I/II clinical trial.

  * A Phase I clinical trial tests the safety and toxicity of adding an investigational device NovoTTF-200A to standard-of-care drug Pembrolizumab to use for further studies.
  * A Phase II clinical trial tests how well the combination works for your brain disease. "Investigational" means that the device is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved NovoTTF-200A for your brain metastasis from melanoma.

A metastatic brain tumor is usually found when a cancer patient begins to experience neurological symptoms and a brain scan (CT or MRI) is ordered. However, some participants are symptom-free and are only diagnosed with brain metastases with MRI or CT scans for another reason.

The NovoTTF-200A System is a portable device which produces changing electrical fields, called Tumor Treatment Fields ("TTFields") within the human body. TTFields stop the growth of tumor cells resulting in cell death of the rapidly dividing cancer cells. TTFields may also sensitize the tumor cells to immune therapies and this is the rationale for combining NovoTTF-200A and Pembrolizumab.

The system is a portable, light-weighted, battery operated device designed to deliver TTFields directly to the region where brain metastasis are. The device can be carried backpack while working or doing other activities of daily living.

ELIGIBILITY:
Subject Inclusion Criteria

* For phase 1 portion: Participants must have histologically confirmed melanoma (either measurable or evaluable) that is metastatic to the brain (TNM classification: Any T, Any N and M1d with or without M1a or M1b involvement). Direct pathological confirmation of metastatic melanoma from the brain is not necessary, provided that the lesions on neuroimaging (either gadolinium-enhanced MRI (preferred) or contrast-enhanced CT of the head) possess typical characteristics of brain metastases as determined by the treating investigator. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm by MRI. Evaluable lesions are those that are <10 mm in all dimensions. Both BRAF wild-type and mutated melanomas are eligible; BRAF mutated patients are required to have previously progressed on or not tolerate BRAF/MEK targeted therapy.
* For phase 2 portion: Participants must have histologically confirmed and measurable melanoma tumor that is metastatic to the brain (TNM classification: Any T, Any N and M1d with or without M1a or M1b involvement). Direct pathological confirmation of metastatic melanoma from the brain is not necessary, provided that the lesions on neuroimaging (either gadolinium-enhanced MRI (preferred) or contrast-enhanced CT of the head) possess typical characteristics of brain metastases as determined by the treating investigator. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm by MRI. Both BRAF wild-type and mutated melanomas are eligible; BRAF mutated patients are required to have previously progressed on or not tolerate BRAF/MEK targeted therapy.
* Age 18 or above.
* ECOG performance status 0-1 or Karnofsky ≥80 (see Appendix A)
* Life expectancy of greater than 6 months.
* Participants must have normal organ and marrow function as defined below

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 x institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * albumin >2.5 mg/dL
  * INR or PT ≤1.5 x ULN unless subject is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
  * aPTT ≤1.5 x ULN unless subject is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Have either measurable or evaluable disease in Phase I & must have measurable disease in Phase II based on the RANO criteria for brain metastases (maximum tumor diameter is 3 cm).
* Have at least 1 untreated brain metastasis for response assessment. Subjects with solitary melanoma brain metastasis should not be treated with either surgery or radiation prior to trial entry.
* Confirm available archival or newly obtained tissue (either brain or systemic) from prior core or excisional biopsy of a tumor lesion.
* Be willing to comply with NovoTTF-200A device treatment for at least 75% of the time.
* Must have caregiver or support available to assist transducer array exchange.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 14 days (or within 72 hours if deemed necessary by the treating investigator) prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, use barrier methods of contraception, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.8). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception, including spermicide, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* The effects of NovoTTF-200A and pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of administration.
* Ability to understand and the willingness to sign a written informed consent document.

Subject Exclusion Criteria

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to first dose of treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. Subjects with newly diagnosed brain metastasis during checkpoint inhibitor treatment are eligible, as long as they have stable or regressing systemic melanoma and the only site of relapse is in the brain.
* Participants who are receiving any other investigational agents.
* History of hypersensitivity to pembrolizumab or any of its excipients.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women, or those expecting to conceive or father children within the projected duration of the trial (starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment), are excluded from this study.
* A diagnosis of immunodeficiency or HIV.
* A known history of active TB (Bacillus Tuberculosis)
* Systemic steroid therapy at a dose equivalent to 4 mg daily of dexamethasone or more, or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Hypersensitivity to hydrogel.
* Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to the agents.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Known leptomeningeal metastasis. Confirmation of negative leptomeningeal metastasis, either by CSF analysis or by neuroimaging staging (no leptomeningeal enhancement or drop metastasis on gadolinium-enhanced head or total spine MRI, respectively) should be determined by the treating investigator. However, it is recommended that both CSF and neuroimaging be obtained because both modalities have limitations in sensitivity and specificity.

Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of enlarging brain metastases, and are not using excessive steroids (defined as a dexamethasone dose of >4 mg daily or equivalent) for at least 7 days prior to trial treatment. This exception does not include leptomeningeal metastasis, which is excluded regardless of clinical stability.

* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Pre-existing hypothyroidism and type I diabetes mellitus (including those from prior anti-cancer monoclonal antibody treatment) are not considered as active autoimmune diseases. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Subject who received a live vaccine within 30 days of planned start of study therapy.
* Implanted pacemaker, defibrillator, deep brain stimulator, or documented clinically significant arrhythmias.
* Evidence of increased intracranial pressure meets any of the follow criteria of raised intracranial pressure:
* midline shift >5mm
* clinically significant papilledema
* nausea/vomiting related to raised intracranial pressure
* reduced level of consciousness related to raised intracranial pressure
* Subjects who received major surgery have not recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity | 21 Days
  Dose limited toxicity is considered grade 3 or higher treatment-related adverse events.

SECONDARY OUTCOMES:
Overall Response Rate | defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive up to 100 months
12-month Overall Survival Rate | 1 Year after last study treatment
  Kaplan-Meir estimates
6-month progression-free survival (PFS) rate | 6 months after last study treatment
  Kaplan-Meir estimates
Quality of Life Assessment | Baseline, 63 Days, 129 Days, 189 Days, 30 days after last study treatment
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) has been used extensively in many cancer clinical trials and it is supplemented by the EORTC QLQ Brain Neoplasm 20 (BN20), which was developed specifically for patients with brain cancer.
  The EORTC QLQ-C30 consists of 30 items and the measurement ranges from 0 to 100, with higher score meaning better outcome in the Global Health Status domain but worse outcomes in the Functional and Symptom Scales.
  The EORTC QLQ-BN20 consists of 20 items and the measurement ranges from 0 to 100, with higher score meaning worse outcome in 4 scales (future uncertainty, visual disorder, motor dysfunction and communication deficit) and 7 individual items (headache, seizure, drowsiness, hair loss, itchy skin, weakness of legs and bladder control).

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Wong, MD, Principal Investigator — Lifespan Cancer Institute
Locations (1):
- Lifespan Cancer Institute, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No